CLINICAL TRIAL: NCT00006313
Title: Hormone Therapy Effects on CVD Risk Factors
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 921; R03HL062429 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2002-09

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To conduct extended analysis of the Postmenopausal Estrogen/Progestins Intervention PEPI trial database to address questions related to cardiovascular disease risk factor response and the possible determinants of this response.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease is the leading cause of death among postmenopausal women. Growing evidence exists that hormone replacement therapy (HRT) may reduce cardiovascular disease and mortality. This has led to the use of postmenopausal HRT for primary prevention of heart disease, however it remains unresolved which women are likely to benefit most from this clinical approach. This is a complicated question because many potential mechanisms are involved by which hormone therapy (HRT) may confer cardioprotection. The Postmenopausal Estrogen/Progestins Intervention (PEPI) trial examined the relative impact of four regimens of hormone therapy on a range of cardiovascular disease risk factors (e.g. lipids, blood pressure, insulin/glucose, hemostasis factors). The trial was well conducted; its data have been thoroughly edited and have yielded a series of important publications. To date, however, publications have focused on average effects without a thorough exploration of the range of, and interplay among, the various effects across the 875 enrolled in the trial.

DESIGN NARRATIVE:

The study extended the analysis of PEPI data by: 1) characterizing the distributions of responses to hormone therapy with respect to risk factors for cardiovascular disease (lipids/lipoproteins, blood pressure, insulin/glucose, hemostasis factors); 2) examining the multivariate patterns of treatment effects among these cardiovascular risk factors and on other outcomes (symptomatology, bone, endometrial); 3) examining clinical and demographic factors that may affect these relationships and, in doing so, characterizing women who may vary with respect to their "sensitivity" to the separate effects of estrogen and progestin therapy; 4) examining closely patterns of adherence and their relationship to response. An experienced team of statisticians/epidemiologists conducted and planned to publish results from these analyses.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-06; Study Completion 2000-06 (Actual)